CLINICAL TRIAL: NCT01825304
Title: the Study of Using Esophageal Pressure to Guide the PEEP Setting in Abdominal Hypertension Patients Who Undergoing Mechanical Ventilation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Collaborators: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Gang Li, PLA Research Institute of general surgery, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CC110-92
Record Dates: First submitted 2013-04-02; First posted 2013-04-05 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2011-10

CONDITIONS: ARDS; Intra-abdominal Hypertension
Keywords: mechanical ventilation; Intra-abdominal hypertension; positive end-expiratory pressure
MeSH Terms: conditions — Intra-Abdominal Hypertension

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- esophageal pressure ,titrated setting (Active Comparator)
  Interventions: Device: titrated setting peep
- ARDSNet recommendations,peep (Other)
  Interventions: Device: titrated setting peep

INTERVENTIONS:
Device: titrated setting peep — titrated setting peep according to esophageal pressure in experimental group; setting peep on the patient's PaO2 and FiO2 in control group.

SUMMARY:
Intra-abdominal hypertension can increase the pleural pressure, and then end-expiratory transpulmonary pressures will be turn to negative, Pulmonary atelectasis/acute lung injury/acute respiratory distress syndrome will appear. In the group of people who suffering intra-abdominal hypertension, the investigators use the pressure of esophagus to speculate the Intrathoracic pressure, and to setting PEEP in order to decrease the happening of ALI/ARDS, which may decrease morbidity in this population.

ELIGIBILITY:
Inclusion Criteria:

* intra-abdominal hypertension
* mechanical ventilation
* sedation

Exclusion Criteria:

* underlying pulmonary disease
* age older than 60 years and younger than 18 years
* vital signs were not stable
* non voluntary

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
ventilator-free days | 28d
  Comparison of two groups the duration of ventilation-free in 28d,ventilator-free day include weaning from mechanical ventilation more than 24h.

SECONDARY OUTCOMES:
mortality | 28d
  28-Day mortality include patients who giving up treatment due to critical condition

CONTACTS AND LOCATIONS:
Locations (1):
- Ventilator, Bern, Canton of Bern, Switzerland